CLINICAL TRIAL: NCT00049803
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Trial Comparing the Effects of Orally Administered Xyrem (Sodium Oxybate) With Placebo for the Treatment of Narcolepsy
Brief Title: Safety and Efficacy of Xyrem Oral Solution (Sodium Oxybate) Compared With Placebo in Narcoleptic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orphan Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMC-SXB-15
Record Dates: First submitted 2002-11-13; First posted 2002-11-15 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Sodium Oxybate; Cataplexy; Excessive Daytime Sleepiness; GHB; Gamma Hydroxybutyric Acid; Orphan Medical; Orphan Drug
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence | interventions — Sodium Oxybate

INTERVENTIONS:
Drug: sodium oxybate

SUMMARY:
The initial portion of the protocol involves discontinuing any medications for cataplexy that the patient may be taking. Subsequently, the patient is prescribed a dose of oral solution of study drug or placebo over a 10-11 week period. During the trial, narcolepsy symptoms will be evaluated. Participants are allowed to continue using stimulant medications at constant doses during the study. A total of 1 to 3 daytime visits in addition to 4 overnight visits to the sleep center will be required to complete the study.

ELIGIBILITY:
INCLUSION CRITERIA

* Have signed & dated informed consent before beginning protocol procedures.
* Willing & able to complete entire trial as described in protocol.
* 16 years of age or older.
* Have a history and presenting symptoms of excessive daytime sleepiness.
* Have a history of cataplexy localizable to a specific muscle group(s) or part(s) of body during which the patient is lucid (not experiencing an inadvertent nap or micro sleep).
* Have valid PSG & MSLT scores (collected during an overnight test) within last five years and a current diagnosis of narcolepsy according to the following criteria established by the American Sleep Disorders Association: (1) Recurrent daytime naps or lapses into sleep occur almost daily for at least 3 months; (2) Sudden bilateral loss of postural muscle tone occurs in association with intense emotion (cataplexy); (3) Polysomnography demonstrates one or more of the following: (a) Sleep latency less than 10 minutes; (b) REM sleep latency less than 20 minutes; (c) An MSLT that demonstrates a mean sleep latency of less than 5 minutes; (d) Two or more sleep-onset REM periods
* Females who are surgically sterile, two years post-menopausal, or if of child-bearing potential, using a medically accepted method of birth control and agree to continue use of this method for the duration of the trial.
* In the opinion of the investigator, have adequate support for the duration of trial to include transportation to and from trial site. In addition, if in the investigator's assessment it is clinically indicated, the patient is willing to not operate a car or heavy machinery for the duration of the trial or for as long as the investigator deems clinically indicated.

EXCLUSION CRITERIA

* Received gamma-hydroxybutyrate in the last 30 days.
* Have taken any investigational therapy within 30-day period prior to initial screening visit for this trial.
* Patients taking fluoxetine (Prozac).
* Have been diagnosed with sleep apnea syndrome, defined as an Apnea Index > 10 per hour or an Apnea Hypopnea Index greater than 15 per hour, or have any other cause of daytime sleepiness, and have any other disorder(s) that can be considered a primary cause of excessive daytime sleepiness.
* Taking hypnotics, tranquilizers, antihistamines (except for non-sedating antihistamines), benzodiazepines or clonidine at the start of the baseline period. Patients taking anticonvulsants are not eligible to participate even if willing to washout anticonvulsants for the trial.
* Experiencing unstable cardiovascular, endocrine, neoplastic (excluding localized basal cell carcinoma), gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurological (other than narcolepsy/cataplexy), pulmonary, and/or renal disease which would place the patient at risk during the trial or compromise objectives outlined in the protocol.
* Have psychiatric disorders, major affective or psychotic disorders, or other problems that, in the investigator's opinion, would preclude the patient's participation and completion of this trial or compromise reliable representation of subjective symptoms.
* Have current or recent (within one year) history of a substance use disorder including alcohol abuse as defined by DSM-IV.
* Serum creatinine greater than 2.0 mg/dL, abnormal liver function tests (SGOT [AST] or SGPT [ALT] more than twice the upper limit of normal), or elevated serum bilirubin (more than 1.5 times upper limit of normal), or pre-trial ECG results demonstrating clinically significant arrhythmias, greater than a first degree AV block or a history of myocardial infarction within last six months.
* Have an occupation that requires variable shift work or routine night shift.
* Have a clinically significant history of seizure disorder, a history of clinically significant head trauma (i.e., concussion resulting in clinically significant loss of consciousness) or past invasive intracranial surgery, and are taking anticonvulsant medications.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2000-12; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: William Houghton, MD, Study Chair — Orphan Medical; Harry N Cook, MBA, RPh, Study Director — Orphan Medical
Locations (44):
- United States (36):
  - Sleep Disorders Center of Alabama, Inc., Birmingham, Alabama
  - Pacific Sleep Medicine Services, La Jolla, California
  - Stanford Sleep Disorders Clinic, Stanford, California
  - St. Petersburg Sleep Disorders Center, St. Petersburg, Florida
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Sleep Disorders Center--Division of Neurology, Evanston, Illinois
  - Peoria Pulmonary Associates, Ltd., Peoria, Illinois
  - The Center for Sleep and Wake Disorders/Midwest Neurology, Danville, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Chest Medicine Associates DBA/Sleep Medicine Specialists, Louisville, Kentucky
  - LSU Health Science Center, Shreveport, Louisiana
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Center for Sleep Diagnostics, Newton, Massachusetts
  - Department of Neurology, Worcester, Massachusetts
  - Washington University -- Sleep Medicine Center, St Louis, Missouri
  - Sleep/Wake Center 7N2 -- Bellevue Hospital Center, New York, New York
  - The Sleep Center - Community General Hospital, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Central Carolina Neurology & Sleep, Salisbury, North Carolina
  - CSC Research -- Grove City Sleep Diagnostic Center, Grove City, Ohio
  - Southwest Cleveland Sleep Center, Middleburg Heights, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Pharmaceutical Trials, Inc., Tulsa, Oklahoma
  - Rhode Island Hospital - Division of Pulmonary, Sleep and Critical Care Medicine, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Charleston Pulmonary Associates PA, Charleston, South Carolina
  - Low Country Lung and Critical Care PA, Charleston, South Carolina
  - Palmetto Baptist Medical Center Sleep Disorders Center, Columbia, South Carolina
  - Charleston Pulmonary Associates PA, Mt. Pleasant, South Carolina
  - Sleep Medicine Assoc PLLC -- Summit Medical Center, Hermitage, Tennessee
  - The Houston Sleep Center, Houston, Texas
  - Sleep Medicine Associates of Texas, Plano, Texas
  - Sleep Disorders Center -- Eastern Virginia Medical School -- Sentara General Hospital, Norfolk, Virginia
  - VCU Health System MCV Hospitals - Sleep Disorders Center, Richmond, Virginia
  - Swedish Sleep Medicine Institute, Seattle, Washington
- Canada (7):
  - Canadian Sleep Institute, Calgary, Alberta
  - Vancouver Hospital -- Sleep Disorders Clinic, Vancouver, British Columbia
  - Saint John Regional Hospital -- Somnology Program, Saint John, New Brunswick
  - The Ottawa Hospital Sleep Centre -- Ottawa Hospital -- Civic Campus -- Sleep Laboratory, Ottawa, Ontario
  - The Sleep Disorders Clinic of the Centre for Sleep and Chronobiology, Toronto, Ontario
  - Brain & Sleep Diagnostic Center, Toronto, Ontario
  - Sleep Disorder Centre -- Hopital du Sacre-Coeur, Montreal, Quebec
- Neurologische Poliklinik - Universitats Spital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] A randomized, double blind, placebo-controlled multicenter trial comparing the effects of three doses of orally administered sodium oxybate with placebo for the treatment of narcolepsy. Sleep. 2002 Feb 1;25(1):42-9. PMID 11833860
- [Background] Scrima L, Hartman PG, Johnson FH Jr, Thomas EE, Hiller FC. The effects of gamma-hydroxybutyrate on the sleep of narcolepsy patients: a double-blind study. Sleep. 1990 Dec;13(6):479-90. doi: 10.1093/sleep/13.6.479. PMID 2281247
- [Background] Lammers GJ, Arends J, Declerck AC, Ferrari MD, Schouwink G, Troost J. Gammahydroxybutyrate and narcolepsy: a double-blind placebo-controlled study. Sleep. 1993 Apr;16(3):216-20. doi: 10.1093/sleep/16.3.216. PMID 8506453
- [Background] A 12-month, open-label, multicenter extension trial of orally administered sodium oxybate for the treatment of narcolepsy. Sleep. 2003 Feb 1;26(1):31-5. PMID 12627729
- [Derived] Husain AM, Bujanover S, Ryan R, Scheckner B, Black J, Profant J. Incidence and duration of common, early-onset adverse events occurring during 2 randomized, placebo-controlled, phase 3 studies of sodium oxybate in participants with narcolepsy. J Clin Sleep Med. 2020 Sep 15;16(9):1469-1474. doi: 10.5664/jcsm.8530. PMID 32356515
- [Derived] Roth T, Dauvilliers Y, Guinta D, Alvarez-Horine S, Dynin E, Black J. Effect of sodium oxybate on disrupted nighttime sleep in patients with narcolepsy. J Sleep Res. 2017 Aug;26(4):407-414. doi: 10.1111/jsr.12468. Epub 2016 Nov 3. PMID 27807903
- [Derived] Bogan R, Swick T, Mamelak M, Kovacevic-Ristanovic R, Lai C, Black J, Villa KF, Montplaisir J. Evaluation of Quality of Life in Patients With Narcolepsy Treated With Sodium Oxybate: Use of the 36-Item Short-Form Health Survey in a Clinical Trial. Neurol Ther. 2016 Dec;5(2):203-213. doi: 10.1007/s40120-016-0053-5. Epub 2016 Oct 24. PMID 27778193